CLINICAL TRIAL: NCT03713931
Title: BUSQUEDA ACTIVA DE CASOS DE EPOC EN EL PRIMER NIVEL DE ATENCION: USO DEL SCORE PUMA PARA TAMIZAJE DE EPOC
Brief Title: PUMA Implementation 2
Acronym: IPUMA2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gustavo Zabert, MD (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Gustavo Zabert, MD, Professor, MD, Asociacion Latinoamericana de Torax
Organization: Asociacion Latinoamericana de Torax (Industry)
Other Study IDs: IPUMA002
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Adult; Risk Factors; Primary Care; COPD; Screening Score; Spirometry; Diagnosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease | interventions — Spirometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PUMA Score questionnaire — Every patient who meet the criteria for active search (older than 40 years, smokers or ex-smokers of more than 10 pack-years who attend the usual care in the first level of care) will be scored with the PUMA´s questionnaire in an application and electronic database (RedCap) specially designed for the active search of cases.
  Patients with PUMA´s score ≥ 5, and without exclusion criteria for spirometry will be referred to perform spirometry at the institution
  Other Names: Spirometry

SUMMARY:
COPD is underdiagnosed and spirometry is not widely available in primary care settings. This study explore the value of PUMA´s questionnaire in a case finding strategy to detect patients to perform spirometry in a real world scenario of primary care health venues.

DETAILED DESCRIPTION:
PUMA (Prevalence StUdy and Regular Practice, Diagnosis and TreatMent, Among General Practitioners in Populations at Risk of COPD in Latin America) study, a multicenter, multinational, cross-sectional, non-interventionist study, explored COPD prevalence among high risk patients assisted in primary care centers in 4 Latin American countries High risk condition was defined if the patient was older than 40 years and current or former smokers (≥10 pack-years, ≥50 pipes/year, or ≥50 cigars/year), and/or reported exposure to biomass smoke, such as wood or coal, for cooking or heating (exposure ≥100h/year). Patients were enrolled during routine, spontaneous or scheduled visits to their medical appointment neither related with the study nor respiratory services or specialists as well. COPD was defined as post-bronchodilator (post-BD) forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) <0.70 and the lower limit of normal (LLN) of FEV1/FVC.

Based on PUMA study data, a simple and a weighted score was constructed with seven variables: sex, age, pack-years smoking, dyspnea, sputum, cough and previous spirometry selected from the PLATINO questionnaire. The score had a mean accuracy for detecting COPD (post-BD FEV1/FVC <0.70) for high risk population of 76% and 79% for the simple and weighted scores, respectively.

This study is a prospective case finding study based on PUMA score as screening tool in unselected high risk patients attending to a primary care health care venue in real world scenario (e.g. community hospital, university institutions or other primary care settings). Patients older than 40 years of age and ever smoker of at least 10 pack year will be asked to complete the PUMA questionnaire through an specially designed application and electronic database (RedCap). All patients who with PUMA score ≥ 5, will be referred to perform spirometry at the institution.

Recruitment will be done by primary care physicians during regular consultations for any reason and spirometry will be performed by qualified technicians using the EasyOne® (nnd) spirometer. The quality of the spirometry will be evaluated by the central team that may request a second measurement to satisfy quality.

COPD will be diagnosed with fixed FEV1/FVC ratio (forced expiratory volume in the first second or FEV1 divided by forced vital capacity or FVC) less than 0.7.

Results will be reported to the primary care doctor and the patient

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who attend the first level of care for any reason in usual care
* Informed consent: subjects must give their signed and dated informed consent to participate.
* Age older 40 years of age
* Smoker or ex-smoker of more than 10 years package

Exclusion Criteria:

* pregnancy,
* patients with contraindication for spirometry (thoracic, abdominal or neurological surgery,
* acute coronary syndrome, retinal detachment, hospitalization for any cardiac problem in the last 3 months)
* patients who at the time of performing the spirometry heart rate ≥ 120 bpm,
* patients with physical or mental incapacity to answer the questionnaire
* patients with physical or mental disability complete the study procedures,
* patients being treated for tuberculosis or any other infectious respiratory disease
* current participants of a clinical trial.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this active case finding study will be patients older than 40 years old, smokers or ever-smokers of more than 10 pack-years, who attend to the first level of care in the real world scenario of primary care facilities (for example: community hospital, university institutions or other environments) without respiratory specialists.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2018-12-21 (Estimated); Study Completion 2019-01-21 (Estimated)

PRIMARY OUTCOMES:
COPD prevalence | 2 days
  FEV1 / FVC post-BD <0.70

SECONDARY OUTCOMES:
PUMA ≥ 5 prevalence | 1 day
  cases with PUMA´s score ≥ 5

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo E Zabert, MD, Principal Investigator — ALAT; Ignacio Zabert, MD, Study Director — ALAT; Fabian Mariluan, MD, Study Director — ALAT
Locations (5):
- Argentina (5):
  - Sistema Integrado de Salud, Tandil, Buenos Aires
  - Hospital Perrando, Resistencia, Chaco Province
  - Hospital "V Sanguinetti", Comodoro Rivadavia, Chubut Province
  - CEPROSS, San Salvador, Entre Ríos Province
  - Hospital Alfredo Metraux,, Maipú, Mendoza Province

IPD SHARING:
Plan to Share IPD: Yes
Questionnaire and spirometric data will be available for review and analysis
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 month after last patient recruited
Access Criteria: IPD will be shared with other research groups interested in similar initiatives. Information about proyect and responsable investigator/person will be requested. Each requests will be reviewed by PUMA 2 team and ALAT reserach board

REFERENCES:
- [Result] Buist AS, McBurnie MA, Vollmer WM, Gillespie S, Burney P, Mannino DM, Menezes AM, Sullivan SD, Lee TA, Weiss KB, Jensen RL, Marks GB, Gulsvik A, Nizankowska-Mogilnicka E; BOLD Collaborative Research Group. International variation in the prevalence of COPD (the BOLD Study): a population-based prevalence study. Lancet. 2007 Sep 1;370(9589):741-50. doi: 10.1016/S0140-6736(07)61377-4. PMID 17765523
- [Result] Menezes AM, Perez-Padilla R, Jardim JR, Muino A, Lopez MV, Valdivia G, Montes de Oca M, Talamo C, Hallal PC, Victora CG; PLATINO Team. Chronic obstructive pulmonary disease in five Latin American cities (the PLATINO study): a prevalence study. Lancet. 2005 Nov 26;366(9500):1875-81. doi: 10.1016/S0140-6736(05)67632-5. PMID 16310554
- [Result] Caballero A, Torres-Duque CA, Jaramillo C, Bolivar F, Sanabria F, Osorio P, Orduz C, Guevara DP, Maldonado D. Prevalence of COPD in five Colombian cities situated at low, medium, and high altitude (PREPOCOL study). Chest. 2008 Feb;133(2):343-9. doi: 10.1378/chest.07-1361. Epub 2007 Oct 20. PMID 17951621
- [Result] Echazarreta AL, Arias SJ, Del Olmo R, Giugno ER, Colodenco FD, Arce SC, Bossio JC, Armando G, Soriano JB; Grupo de estudio EPOC.AR. Prevalence of COPD in 6 Urban Clusters in Argentina: The EPOC.AR Study. Arch Bronconeumol (Engl Ed). 2018 May;54(5):260-269. doi: 10.1016/j.arbres.2017.09.018. Epub 2017 Dec 6. English, Spanish. PMID 29221827
- [Result] Sobrino E, Irazola VE, Gutierrez L, Chen CS, Lanas F, Calandrelli M, Ponzo J, Mores N, Seron P, Lee A, He J, Rubinstein AL. Estimating prevalence of chronic obstructive pulmonary disease in the Southern Cone of Latin America: how different spirometric criteria may affect disease burden and health policies. BMC Pulm Med. 2017 Dec 11;17(1):187. doi: 10.1186/s12890-017-0537-9. PMID 29228947
- [Result] Schiavi E, Stirbulov R, Hernandez Vecino R, Mercurio S, Di Boscio V; Puma Team. COPD screening in primary care in four Latin American countries: methodology of the PUMA Study. Arch Bronconeumol. 2014 Nov;50(11):469-74. doi: 10.1016/j.arbres.2014.03.006. Epub 2014 May 9. English, Spanish. PMID 24816036
- [Result] Bergna MA, Garcia GR, Alchapar R, Altieri H, Casas JC, Larrateguy L, Nannini LJ, Pascansky D, Grabre P, Zabert G, Miravitlles M. Development of a simple binary response questionnaire to identify airflow obstruction in a smoking population in Argentina. Eur Respir Rev. 2015 Jun;24(136):320-6. doi: 10.1183/16000617.00005214. PMID 26028643
- [Result] Laniado-Laborin R, Rendon A, Bauerle O. Chronic obstructive pulmonary disease case finding in Mexico in an at-risk population. Int J Tuberc Lung Dis. 2011 Jun;15(6):818-23. doi: 10.5588/ijtld.10.0546. PMID 21575305
- [Result] Lopez Varela MV, Montes de Oca M, Rey A, Casas A, Stirbulov R, Di Boscio V; PUMA Team. Development of a simple screening tool for opportunistic COPD case finding in primary care in Latin America: The PUMA study. Respirology. 2016 Oct;21(7):1227-34. doi: 10.1111/resp.12834. Epub 2016 Jun 20. PMID 27319305
- [Result] Stanley AJ, Hasan I, Crockett AJ, van Schayck OC, Zwar NA. Validation of the COPD Diagnostic Questionnaire in an Australian general practice cohort: a cross-sectional study. Prim Care Respir J. 2014 Mar;23(1):92-7. doi: 10.4104/pcrj.2014.00015. PMID 24570082
- [Result] Price DB, Tinkelman DG, Nordyke RJ, Isonaka S, Halbert RJ; COPD Questionnaire Study Group. Scoring system and clinical application of COPD diagnostic questionnaires. Chest. 2006 Jun;129(6):1531-9. doi: 10.1378/chest.129.6.1531. PMID 16778271